CLINICAL TRIAL: NCT01329237
Title: Comparison of the Everolimus Eluting (XIENCE-V® or PROMUS® Stent) With the Biolimus A9 Eluting NOBORI® Stent in All-comers: a Randomized Open Label Study The COMPARE II Trial Imaging and Vasomotion Substudy
Brief Title: COMPARE-II- Vasomotion and Imaging Substudy
Acronym: COMPARE-IT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Freiburg (Other)
Responsible Party: TOGNI Mario/Professor of Medicine, University of Fribourg Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COMPARE-II-Imaging
Record Dates: First submitted 2011-03-28; First posted 2011-04-05 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-01

CONDITIONS: Coronary Artery Disease
Keywords: drug-eluting stent; coronary endothelial function; coronary imaging
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dynamic physical exercise OCT (Other): dynamic physical exercise and optical coherence tomography imaging
  Interventions: Other: dynamic physical exercise and OCT imaging

INTERVENTIONS:
Other: dynamic physical exercise and OCT imaging — supine dynamic physical exercise during coronary angiography and optical coherence tomography OCT imaging of the coronary stent

SUMMARY:
The purpose of the study is to compare strut coverage and neointimal thickness between everolimus eluting (XIENCE-V® or PROMUS® stent) and biolimus A9 eluting NOBORI Stent 14 months after stent implantation and to determine the coronary endothelial function after everolimus eluting (XIENCE-V® or PROMUS® stent) and biolimus A9 eluting NOBORI Stent 14 months after stent implantation by using supine bicycle exercise testing to assess coronary vasomotor response to exercise.

DETAILED DESCRIPTION:
DESIGN:

Imaging and vasomotion Substudy:

50 consecutive patients enrolled in the COMPARE II trial at the University of Fribourg Medical Center will undergo follow-up re-angiography 14 months after index procedure with assessment of Optical coherence tomography (OCT) and vasomotion testing.

ENDPOINT SUBSTUDY (all at 14 months):

Primary endpoint imaging: percentage of uncovered stent struts per lesion and mean neointimal thickness assessed by OCT.

vasomotion: coronary vasomotion assessed with quantitative coronary angiography at rest and during supine bicycle exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patient enrolled in the COMPARE II trial with successful stent implantation and absence of binary restenosis or severe progression of coronary artery disease at 14 months follow-up.
* Patient consent to undergo a non-scheduled follow- up angiography with imaging study and bicycle exercise testing

Exclusion Criteria:

1. Inability to provide informed consent
2. Inability to perform a supine bicycle exercise stress test
3. Binary in stent restenosis of the target vessel
4. Acute Coronary Syndrome, Acute Myocardial Infarction
5. Patients with stent thrombosis following the index procedure
6. Female of childbearing potential ( age ≤ 50 years and last menstruation within the last 12 months ), who did not undergo tubal ligation, ovariectomy or hysterectomy
7. Known intolerance to heparin, contrast material
8. History of bleeding diathesis or known coagulopathy
9. Age ≥ 80 years
10. Hemodynamic instability
11. Renal failure (creatinine clearance ≤ 40 ml/min)
12. OCT / IVUS technically not feasible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
percentage of uncovered stent struts per lesion assessed by OCT | within 14 months after percutaneous coronary stent implantation

SECONDARY OUTCOMES:
coronary vasomotor function | within 14 months after stentimplantation
  coronary vasomotion assessed with quantitative coronary angiography at rest and during supine bicycle exercise
mean neointimal thickness assessed by OCT | within 14 months after stent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Mario Togni, MD, Principal Investigator — University of Fribourg, Switzerland; Stéphane Cook, MD, Principal Investigator — University of Fribourg, Switzerland; Jean-Christophe Stauffer, MD, Study Chair — Hopital Cantonal HFR, Fribourg, Switzerland; Jean-Jacques Goy, MD, Study Chair — Hopital Cantonal HFR, Fribourg, Switzerland; Gérard Baeriswyl, MD, Study Chair — Hopital Cantonal HFR, Fribourg, Switzerland; Pieter C Smits, MD, PhD, Principal Investigator — Maasstad Ziekenhuis, Rotterdam, The Netherlands
Locations (1):
- Hopital Cantonal HFR, Fribourg, Canton of Fribourg, Switzerland